CLINICAL TRIAL: NCT01390636
Title: Characterizing Diurnal Glucose Patterns of Individuals With Type 1 Diabetes and Eating Disorders
Brief Title: Type 1 Diabetes and Eating Disorder Diurnal Glucose Patterns
Acronym: REACT5
Status: Terminated | Type: Observational
Why Stopped: The study was a collaboration that could not be effectively run.
Sponsor: HealthPartners Institute (Other)
Collaborators: Park Nicollet Foundation (Other); Melrose Institute (Unknown); International Diabetes Center at Park Nicollet (Other)
Responsible Party: Sponsor
Other Study IDs: 04126-11-C
Record Dates: First submitted 2011-06-29; First posted 2011-07-11 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2013-08

CONDITIONS: Type I Diabetes Mellitus Without Complication; Eating Disorder
Keywords: Continuous Glucose Monitoring; Type 1 Diabetes and an Eating Disorder; Eating Disorder Only
MeSH Terms: conditions — Feeding and Eating Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED-DMT1 and ED/only: Eating Disorder and Type 1 Diabetes and only an Eating Disorder

SUMMARY:
The purpose of this study is to use data from the Continuous Glucose Monitor (CGM) to determine the degree of variation in glucose levels of individuals with an eating disorder and type 1 diabetes and only an eating disorder.

DETAILED DESCRIPTION:
The specific aims of the proposed research are to:

2.1 Determine the degree of variation in glycemic profiles of individuals with an Eating Disorder and Type 1 Diabetes (ED-DMT1) and an Eating Disorder only (ED/only); and

2.2 Determine the impact of nutritional intake and planned physical activity on glucose profiles of individuals with ED-DMT1 and ED/only.

These aims will be examined by characterizing:

* glucose exposure, as measured by area under the Ambulatory Glucose Profile (AGP) median curve;
* glucose variability, as measured by the AGP inter-quartile range; and
* glucose stability, as measured by change in the AGP median curve.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the ISL unit at Melrose Institute
* Diagnosed with an eating disorder (Anorexia Nervosa, Bulimia Nervosa or Eating Disorder Not Otherwise Specified)

  1. For ED-DMT1 group: Diagnosis of an eating disorder AND diagnosis of type 1 diabetes.
  2. For ED/only group: Diagnosis of an eating disorder AND no history/diagnosis of type 1 or type 2 diabetes.
* Female.
* At least 14 years of age.
* Able to provide informed consent.

  1. If the potential participant's age is at least 18 years she must be able to provide informed consent.
  2. If the potential participant is less than 18 years she must have a parent or guardian able and willing to provide written informed consent on the participant's behalf. In addition, the participant must be willing to sign a consent on her own behalf.
* Participants must be able and willing to utilize the CGM system and perform required calibrations using self-monitored blood glucose.

Exclusion Criteria:

* Male.
* Age < 14 years.
* History of self-injurious behavior that the senior clinician feels precludes participation.
* Unable to understand the study protocol.
* Unwilling to follow the study protocol.
* Participation in any competing research study.
* Planned ISL admission for <4 days.
* Pregnant.
* Not able to communicate in English.
* Regular use of acetaminophen or acetaminophen containing medications and not able to modify their medication to a non-acetaminophen based medication.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Current Melrose Institute Patient
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Variation in Glycemic Profiles of ED-DMT1 and ED/only | 10 days
  Determine the degree of variation in glycemic profiles of individuals with ED-DMT1 and ED/only using Continuous Glucose Monitoring (CGM). CGM will be graphically and statistically represented by an Ambulatory Glucose Profile (AGP).

SECONDARY OUTCOMES:
Impact of Dietary Intake on Glucose Profiles of ED-DMT1 and ED/only | 10 days
  Determine the impact of dietary intake and planned physical activity on glucose profiles of individuals with ED-DMT1 and ED/only using Continuous Glucose Monitoring (CGM). CGM will be graphically and statistically represented by an Ambulatory Glucose Profile (AGP).

CONTACTS AND LOCATIONS:
Overall Officials: Mazze S Mazze, PhD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- Melrose Institute, Minneapolis, Minnesota, United States